CLINICAL TRIAL: NCT05414968
Title: A Novel Non-Pharmacological Treatment of Diabetic Neuropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Auburn University (Other)
Responsible Party: Principal Investigator, Chad Rose, Assistant Professor, Auburn University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 22-114
Record Dates: First submitted 2022-06-07; First posted 2022-06-10 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: nonpharmacological intervention

STUDY DESIGN:
Intervention Model Description: 16 participants will be recruited (8 pre-neuropathic, 8 neuropathic) to evaluate device feasibility through 10 sessions spread over 14 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pilot Feasibility Arm (Experimental): Each participant will receive the same 45-minute intervention on 10 days spread over no more than 14 days total. At the end of each session, pain will be assessed on scales such as the Defense and Veterans Pain Rating Scale (DVPRS) to establish the safety and feasibility of the proposed intervention.
  Interventions: Device: Non-pharmacological Heat, Pressure, and Vibration

INTERVENTIONS:
Device: Non-pharmacological Heat, Pressure, and Vibration — The innovation central to this approach is in the multifactorial combination of pressure, heat, and vibration stimuli to improve foot sensation. The heat stimuli will be provided with commercially available heating elements. The pressure stimuli will be provided via pneumatic garment. Lastly, the vibrotactile stimuli will be provided with commercially available vibrotactile motors. The non-pharmacological DPN device will be able to safely and consistently control temperature to 100-105°F within 1°F, control pressure to 50 mmHg within 5 mmHg at 0.25 Hz, and provide 5 distinguishable vibrational stimuli to 5 zones on the leg and foot.

SUMMARY:
The objective of the proposed work is to develop non-pharmacological interventions for diabetic peripheral neuropathy (DPN), to improve quality of life of individuals with diabetes, and reduce the prevalence of opiate prescription, sensation loss, falls, and deaths caused by DPN. To this end, the proposed study will investigate and determine the feasibility of the non-pharmacological intervention device. The feasibility study involves 16 participants, split evenly between pre-neuropathic diabetic and neuropathic diabetic participants. During the study, each group will receive the same 45-minute intervention on 10 days spread over no more than 14 days total. Feasibility will be determined by change in pain assessed before and after intervention.

DETAILED DESCRIPTION:
To address a gap in DPN treatments, we propose a pragmatic approach towards the development of mechanistically justified therapies to treat DPN. Specifically, we seek to explore undertested non-pharmacological approaches to DPN management through a pilot study establishing safety and feasibility as quantified by biomechanical and sensory-perception changes.

The innovation central to this approach is in the multifactorial combination of pressure, heat, and vibration stimuli to improve foot sensation by 1) reducing edema in the foot and leg via improved venous return and lymphatic return, 2) improving arterial flow both in large, small, and micro-vascular vessels, 3) stimulating endothelial mechanisms like the increase of nitrous oxide that increases microvascular health through alternating compressive pressures from the foot to the thigh, and 4) stimulating nerves through vibration to facilitate nerve repair. This approach has the potential to address an unmet need in DPN, namely, interventions that can address underlying causes of neuropathy. To this end, the proposed research has two specific aims: 1) the construction of a device capable of applying pressure, heat, and vibration to the entire lower extremity for treatment of neuropathy and 2) validation of safety and feasibility of the non-pharmacological intervention device.

At the beginning of the study, foot sensation and blood flow baseline measures will be taken with the foot sensation diagnostic tool and phase-contrast MRI with a foot/ankle coil (Siemens Foot/Ankle 16) at the Auburn University MRI Research Center, respectively. The foot sensation diagnostic tool has undergone testing with over 100 participants with diabetes, and has shown the ability to establish the threshold sensitivity of the sole of the foot from 0.5 to 10 grams force, an order of magnitude more accurate than the standard clinical monofilament-based measure used to establish foot sensitivity and diagnose DPN. The phase-contrast MRI is a highly accurate measure of blood flow, which we will use to validate the mechanistic hypothesis of the proposed non-pharmacological intervention. The phase-contrast MRI does not require the use of contrast-enhancing dyes, and will therefore exclude fewer diabetic participants than contrast-enhanced MRI scans.

During the study, each participant will receive the same 45-minute intervention on 10 days spread over no more than 14 days total, in a similar manner to IPC studies. At the end of each session, pain will be assessed on scales such as the Defense and Veterans Pain Rating Scale (DVPRS) to establish the safety of the proposed intervention. Feasibility will be determined of time to set up, put on, and take off the device. Pre-study baseline measurements of foot sensation via the assessment tool will be compared to post-study measurements to establish any beneficial effect and provide variance for a power analysis to guide the design of future studies. We hypothesize that non-neuropathic diabetic participants may have subclinical neuropathic symptoms which cannot be measured by standard clinical tools but can be measured by the diagnostic device, which may identify the potential for the device to have preventative as well as treatment applications.

Sample Size Justification: A sample size of 16 subjects (8 with non-neuropathic diabetic and 8 with neuropathic diabetic participants) achieves 80% power to detect an effect size as measured in the change in pain scores of 0.55 using a paired t-test with a one tailed Type I error rate of 0.10. Examination of each subgroup will also be conducted. A sample size of 8 subjects achieves 80% power to detect an effect size as measured in the change in pain scores of 0.8 using a paired t-test with a one tailed Type I error rate of 0.10. Therefore, this small study will have statistical power to observe medium to large changes in pain rating (or foot sensation or blood flow). However, it must be noted that achieving statistical significance is not the primary objective of a pilot study. The primary objective is to demonstrate feasibility of the trial by initiating a small version of the trail, identifying areas requiring refinement, and collecting preliminary data provides preliminary evidence of intended effect.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of type 2 diabetes for at least 5 years
* lab histories that verify participant's control or lack of blood sugars dating back for a period of 1-5 years

Exclusion Criteria:

* other diseases or impairments that could affect results (vascular disease verified from medical history
* ankle-brachial index (ABI) of 0.9 or less

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Pain Assessment | immediately after each session (up to 30 minutes)
  Defense and Veterans Pain Rating Scale (DVPRS)

CONTACTS AND LOCATIONS:
Overall Officials: Chad G Rose, PhD, Principal Investigator — Auburn University
Locations (1):
- Auburn University, Auburn, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
If requested, final, de-identified research data will be made available for sharing to qualified parties by the PI's, so long as such a request does not compromise intellectual property interests, interfere with publication, invade subject privacy, betray confidentiality, or precede data curation. All logs will be anonymized before storage.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will become available no later than 1 year after conclusion of the study, and for at least three years after the conclusion of the study.
Access Criteria: PI Approval.

REFERENCES:
- [Background] Lotz J, Meier C, Leppert A, Galanski M. Cardiovascular flow measurement with phase-contrast MR imaging: basic facts and implementation. Radiographics. 2002 May-Jun;22(3):651-71. doi: 10.1148/radiographics.22.3.g02ma11651. PMID 12006694
- [Background] Feldman EL, Nave KA, Jensen TS, Bennett DLH. New Horizons in Diabetic Neuropathy: Mechanisms, Bioenergetics, and Pain. Neuron. 2017 Mar 22;93(6):1296-1313. doi: 10.1016/j.neuron.2017.02.005. PMID 28334605
- [Background] Buckenmaier CC 3rd, Galloway KT, Polomano RC, McDuffie M, Kwon N, Gallagher RM. Preliminary validation of the Defense and Veterans Pain Rating Scale (DVPRS) in a military population. Pain Med. 2013 Jan;14(1):110-23. doi: 10.1111/j.1526-4637.2012.01516.x. Epub 2012 Nov 8. PMID 23137169